CLINICAL TRIAL: NCT01778088
Title: A Phase 2a, Multi-Center, Open-Label Study of I-131-CLR1404 in Subjects With Recurrent Glioma
Brief Title: Open-Label Study of I-131-CLR1404 in Subjects With Recurrent Glioma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCL-13-001
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — CLR1404

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group (Other): I-131-CLR1404 Injection
  Interventions: Drug: I-131-CLR1404 Injection

INTERVENTIONS:
Drug: I-131-CLR1404 Injection
  Other Names: 18-(p-[I-131]-iodophenyl)octadecyl phosphocholine

SUMMARY:
The purpose of this study is to determine the recommended dosing of I-131-CLR1404, a radiolabeled therapy compound, for treating subjects with glioma.

Subjects who meet study entry criteria will receive I-131-CLR1404. For each subject, the study will be conducted in three phases, dosimetric, therapy, and follow-up. In the dosimetric phase, subjects will receive one 5 mCi dose of the study drug and undergo whole body imaging on on the day of infusion and on post-infusion days 2, 3, and 7 for assessment of biodistribution and tumor uptake of I-131-CLR1404. If normal and expected biodistribution are demonstrated, the subject will begin the therapy phase. In the therapy phase, the subjects will receive a dose based on body surface area and may receive additional doses if they meet dosing criteria. After the last treatment dose, subjects will enter the follow-up phase and will be followed monthly.

All subjects will be prescribed thyroid protection medication to be taken 24 hours prior to injection of the dosimetric dose, and continuing for 14 days after the administration of the therapy dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade glioblastoma multiforme (GBM)
* Failed prior therapy with Avastin
* Radiologic evidence of tumor progression
* Received at least 45 Gy and no more than 66 Gy prior radiotherapy
* Ambulatory with an ECOG performance status of 0 to 2 (Appendix C)
* 18 years of age or older

Exclusion Criteria:

* Received more than 25% of total bone marrow irradiated, total body or hemi-body irradiation or prior radioisotope therapy (except for benign thyroid disease)
* Prior radiation therapy or chemotherapy within 4 weeks of start of study
* Another active medical condition(s) or organ disease(s) that may compromise subject safety or interfere with safety and/or outcome evaluation of study drug
* Laboratory abnormalities, including but not limited to: WBC < 3000/uL, Absolute neutrophil count < 1500/uL, Platelets < 150,000/uL, Hemoglobin ≤ 9.0 gm/dL, Total bilirubin > 1.5 x upper limit of normal for age, SGOT or SGPT > 3 x upper limit of normal for age if no liver metastases or > 5 x upper limit of normal for age in the presence of liver metastases, Serum creatinine > 1.5 x upper limit of normal for age, 2+ proteinuria or casts indicative of intrinsic renal disease
* Treatment with investigational drug, investigational biologic, or investigational therapeutic device within 28 days of initiating study treatment
* Received prior stem cell transplantation
* Clinically significant cardiac co-morbidities including congestive heart failure (New York Heart Association class III-IV heart disease), left ventricular ejection fraction < 40%, unstable angina pectoris, serious cardiac arrhythmia requiring medication or pacemaker, myocardial infarction within past 6 months
* Concurrent or recent (within 1 month) use of thrombolytic agents, or full-dose anticoagulants (except to maintain patency of preexisting, permanent indwelling IV catheters).
* Uncontrolled hypertension as defined by systolic blood pressure > 150 mm/Hg, diastolic blood pressure > 100 mm/Hg or uncontrolled diabetes that would compromise subject safety or interfere with safety and/or outcome evaluation of study drug
* Major surgery within 4 weeks of enrollment
* Poor venous access and unable to receive study drug into a peripheral venous catheter
* Significant traumatic injury within past 4 weeks
* Ongoing or active infection requiring antibiotics or with fever >38.1º C (>101º F) within 3 days of first scheduled day of dosing
* Receiving concurrent hemodialysis or peritoneal dialysis
* Known positive for HIV, Hepatitis C (active, previously treated or both), or is Hepatitis B core antigen positive
* Pregnant or lactating
* Hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 6-month survival rate of subjects receiving I-131-CLR1404 for relapsed glioma | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Minesh Mehta, M.D., FASTRO, Principal Investigator — University of Marylannd School of Medicine
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States